CLINICAL TRIAL: NCT02536079
Title: NeuroAiD Safe Treatment Registry
Acronym: NeST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHIMES Society (Other)
Collaborators: Moleac Pte Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NeST2014
Record Dates: First submitted 2015-08-26; First posted 2015-08-31 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Brain Injury; NeuroAiD Use
MeSH Terms: conditions — Brain Injuries | interventions — Neuroaid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: NeuroAiD
  Other Names: MLC601; MLC901

SUMMARY:
The NeST registry is a pro-active industry-academic collaboration to assess the use and safety of NeuroAiD in the real world setting. An online entry system was set up to allow easy data entry and retrieval of clinical information.

DETAILED DESCRIPTION:
The NeST Registry is designed as a product registry that would provide information on the use and safety of NeuroAiD in clinical practice. An online NeST Registry was set up to allow easy entry and retrieval of essential information including demographics, medical conditions, clinical assessments of neurological, functional, and cognitive state, compliance, concomitant medications and side effects if any, among patients on NeuroAiD. Participation is voluntary. Data collected are similar to information obtained during standard care and are prospectively entered by the participating physicians at baseline (before initialization of NeuroAiD) and during subsequent visits. The follow up visits are timed with clinical appointments. Anonymized data will be extracted and collectively analyzed. Initial target sample size for the registry is 2000.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Any age
* Taking, or has been prescribed NeuroAiD for any duration as judged by the physician and/or the participant
* Agrees to be included in the registry and allows retrieval and analysis of data in accordance with local requirements

Exclusion Criteria:

* Unwillingness to participate
* Contraindication to NeuroAiD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The NeST Registry is a product-specific and safety outcome registry that includes patients who are taking NeuroAiD. Participation is entirely voluntary and an agreement will be obtained before inclusion. The decision on the use of NeuroAiD should be made following a discussion between participant and physician and only then will the option of participation in the registry be considered.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-06; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing adverse events | 3 months
  Adverse events categorized according to individual events, organ system, severity (mild, moderate, severe), and relatedness (based on WHO-World Health Organization - Uppsala Monitoring System as 'possibly' 'probably' or 'definitely' related)

SECONDARY OUTCOMES:
Functional status based on modified Rankin Scale | 1, 2, 3 months
  0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Neurological status based on Glasgow Coma Scale | 1, 2, 3 months
  to assess level of consciousness: eye opening, Eye opening 4, Eye Opening Response
  * Spontaneous--open with blinking at baseline 4 points
  * To verbal stimuli, command, speech 3 points
  * To pain only (not applied to face) 2 points
  * No response 1 point;Verbal Response
  * Oriented 5 points
  * Confused conversation, but able to answer questions 4 points
  * Inappropriate words 3 points
  * Incomprehensible speech 2 points
  * No response 1 point;Verbal Response
  * Oriented 5 points
  * Confused conversation, but able to answer questions 4 points
  * Inappropriate words 3 points
  * Incomprehensible speech 2 points
  * No response 1 point;Motor Response
  * Obeys commands for movement 6 points
  * Purposeful movement to painful stimulus 5 points
  * Withdraws in response to pain 4 points
  * Flexion in response to pain (decorticate posturing) 3 points
  * Extension response in response to pain (decerebrate rigidity )
Neurological status based on National Institute of Health Stroke Scale | 1, 2, 3 months
  Quantify impairment caused by stroke 0- no stroke, 1-4 Minor stroke, 5-15 Moderate,16-20 Moderate to Severe stroke, 21-42 severe stroke
Cognitive status based on Short Orientation-Memory-Concentration Test | 1, 2, 3 months
  test involves 6 items test -1.what year is it now?2.What month is it now?3.Repeat phrase, about what time is it ? (within one hour),Count backwards 20 to 1,Say months in reversw order,repeat phrase just given,
Cognitive status based on Mini-Mental State Examination (MMSE) | 3, 6,9, 12 months
  Orientation, Registration,Attention and Calculation,Recall, Language, Copying,
Cognitive status based on Alzheimer's Disease Assessment Scale- cognitive subscale (ADAS-cog) | 3, 6, 9, 12 months
  World recall, Naming of objects and fingers,Commands,Constructional Praxis,Ideational Praxis,Orientation, World Recognition,Language,Comprehension of spoken language,Word finding difficulty, Remembering test instructions
Cognitive status based on Montreal Cognitive Assessment (MoCA) | 3, 6, 9, 12 months
  Visio spatial /executive,naming, memory ,attention , language,abstraction, delayed recall
Functional outcome based on Bristol Activities of Daily Living (BADL) | 3, 6, 9, 12
  Preparing Food 3 Eating 3 Preparing Drink 3 Drinking 3 Dressing 3 Hygiene 3 Teeth 3 Bath/Shower 3 Toilet/Commode 3 Transfers 3 Mobility 3 Orientation - Time 3 Orientation - Space 3 Communication 3 Telephone 3 Housework/Gardening 3 Shopping 3 Finances 3 Games/Hobbies 3 Transport 3

OTHER OUTCOMES:
Number of patients complying to prescribed dosage of NeuroAiD | 1, 2, 3 months
  Compliance assessed as "since last visit, taking NeuroAiD..." never, 'rarely,' 'sometimes,' 'often,' 'always.'
Glasgow Outcome Scale Extended (GOS-E) | 1, 2, 3 months, additional visit
  For Traumatic Brain injury cohort:This clinical scale is the most widely used outcome measure after TBI. The extended version is rated from 0 (dead) to 8 (full recovery)
Rivermead Post-Concussion Symptom Questionnaire (RPQ) | 1, 2, 3 months, additional visit
  For Traumatic Brain Injury Cohort. This questionnaire is a simple, 10-item measure of outcome mainly used with patients with mild to moderate head injuries. This questionnaire explores the occurrence of 16 post-concussive symptoms such as headaches, fatigue, and restlessness
Modified Barthel Index | 1, 2, 3 months, additional visit
  For Traumatic Brain Injury cohort. This scale assesses functional disability by quantifying patient performance in 10 activities of daily life (ADLs). This scale measures performance and patient independence with respect to self-care, sphincter management, transfers and locomotion. The score is calculated by summing the response value to each item.

CONTACTS AND LOCATIONS:
Overall Officials: Narayanaswamy Venketasubramanian, FRCP, Study Chair — Raffles Neuroscience Centre, Raffles Hospital, Singapore; Ramesh Kumar, FRCS, Principal Investigator — Department of Neurosurgery, Faculty of Medicine, University Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Malaysia; Lyna Soertidewi, MD, Principal Investigator — Department of Neurology, National Brain Center Hospital, Jakarta, Indonesia
Locations (2):
- National Brain Center Hospital, Jakarta, Indonesia
- University Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Venketasubramanian N, Kumar R, Soertidewi L, Abu Bakar A, Laik C, Gan R. The NeuroAiD Safe Treatment (NeST) Registry: a protocol. BMJ Open. 2015 Nov 13;5(11):e009866. doi: 10.1136/bmjopen-2015-009866. PMID 26567259